CLINICAL TRIAL: NCT01783301
Title: A Phase IV, Open-label 2 Arm Trial to Compare the Efficacy and Safety of a Pre-defined Dose of GONAL-f® Based on Antral Follicle Count [Follicles ≥2mm - <11mm]), or AMH for Ovarian Stimulation in Subjects Undergoing Assisted Reproductive Technology (ART) Treatment.
Brief Title: Anti-Mullerian Hormone (AMH) Versus Antral Follicle Count (AFC) Guided rFSH Dosing Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vietnam National University (Other)
Collaborators: Merck Serono Vietnam (Unknown)
Responsible Party: Principal Investigator, Manh Tuong Ho, Dr, Vietnam National University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11/QD-CGRH-NCKH&DT
Record Dates: First submitted 2013-01-17; First posted 2013-02-04 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: Infertility
Keywords: follicle stimulating hormone; ovarian stimulation; antimullerian hormone; antral follicle count; assisted reproductive technologies
MeSH Terms: conditions — Infertility | interventions — follitropin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antral follicle count (Active Comparator): Start dose of recombinant Follicle-Stimulating Hormone (rFSH) based on AFC guide
  * AFC < 6 on both ovary: 375 IU FSH
  * 6<AFC <=15 on both ovary: 225 IU FSH
  * AFC> 15 on both ovary: 150 IU FSH
  Interventions: Drug: FSH
- Anti-Mullerian Hormone (Active Comparator): Start dose of FSH based on AMH guide
  * AMH < 5 pmol/L or < 0.7ng/ml: 375 IU FSH
  * AMH 5 to < 15 pmol/L or 0.7 to 2.1ng/ml: 225 IU FSH
  * AMH ≥ 15 pmol/L or > 2.1ng/ml: 150 IU FSH
  Interventions: Drug: FSH

INTERVENTIONS:
Drug: FSH
  Other Names: GONAL-f

SUMMARY:
The overall objectives of this trial are to:

* To explore the efficacy and safety of using either antral follicle count (AFC) or anti-Mullerian hormone (AMH) to guide the starting dose of GONAL-f® in ovarian stimulation for Assisted Reproductive Technology (ART).
* To assess the differences in both ovarian response and clinical pregnancy rate between subjects with different AFC and AMH levels undergoing ART.

DETAILED DESCRIPTION:
Trial design

This trial is a prospective, Phase IV 2 arm trial exploring the efficacy and safety of using either AFC or AMH to guide the starting GONAL-f® dose for the stimulation treatment of subjects undergoing ART.

Throughout the trial period and before the start of a routine ART cycle, investigators will propose the trial to their potential subjects. All subjects who agree to participate in the trial must sign a consent form, irrespective of whether or not they ultimately agree to have their dose determined by the study protocol. Eligible subjects will be randomised in blocks of 4 at each site via a computer generated random number list to either the AFC guided arm (control) or the AMH guided arm (treatment). The starting doses of GONAL-f® for each arm will be based on the study algorithms, using AFC or AMH guidance.

The investigator will then enter initiate ovarian stimulation with an individualised GONAL-f® dose for that specific subject. This will be maintained for the first 5 days of stimulation after which the dose can be modified based on investigator decision and in accordance with the site's routine clinical practice.

Trial Population

Female partners of infertile couples requiring Assisted Reproductive Technology (ART) treatment.

Data Analysis and Statistics

The primary end-point proportion of patients with desired number of retrieved oocytes (8-12) will be compared between the 2 arms using the chi -square test. The null hypothesis will be that there is no difference between the 2 arms in primary end-point, with the p level set at p=0.05. The secondary end-points will also be compared between the 2 arms using either the Student's t test or anova test.

ELIGIBILITY:
Inclusion Criteria:

* Starting a treatment with GONAL-f® according to the decision of the investigator and in accordance with the indication and dosing recommendation
* Age < 40 years at the time of GONAL-f® dosing
* BMI < 28 kg/m2
* An early follicular phase (Day 2-4) serum levels of basal FSH ≤12 IU/L measured in the site's own laboratory and taken within 2 months prior to down-regulation start
* Receiving long Gonadotropin-Releasing Hormone (GnRH) agonist protocol (starting on day 21 of preceding cycle until day of hCG)
* Agreement to participate in the study, and to disclose any medical events to the investigator. The subject must be willing and able to comply with the protocol requirements for the duration of the study.
* Have given written informed consent with the understanding that the subject may withdraw consent at any time without prejudice to future medical care.

Exclusion Criteria:

* Simultaneous participation in an interventional clinical trial.
* Concommitant use of either Luteinizing Hormone or human menopausal gonadotropin/urinary FSH preparations in study cycle

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 348 (Actual)
Dates: Start 2011-10; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Number of oocytes retrieved | 30 minutes after oocyte retrieval completed

SECONDARY OUTCOMES:
Symptoms of ovarian hyperstimulation syndrome (OHSS) | in 10 days after hCG injection

CONTACTS AND LOCATIONS:
Overall Officials: Tuong M Ho, MD, Principal Investigator — Vietnam National University HCMC
Locations (1):
- Research Center for Genetics and Reproductive Health, Ho Chi Minh City, Ho Chi Minh, Vietnam